CLINICAL TRIAL: NCT02822092
Title: Striatal Connectivity and Clinical Outcome in Psychosis
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: HS16-0411
Record Dates: First submitted 2016-06-27; First posted 2016-07-04 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Risperidone; Aripiprazole

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Drug Levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with Psychotic Disorders taking Risp. or Arip.: Risperidone or aripiprazole will be administered. Subjects will start risperidone 1 mg qhs or 5mg qhs aripiprazole; on day 4 the daily dose will be increased to 2 mg risperidone or 10mg aripiprazole and to 3 mg risperidone or 15mg aripiprazole at day 7. The target dose is 3 mg risperidone or 15 mg aripiprazole daily but patients who remain psychotic can be increased to 4 mg risperidone or 20mg aripiprazole at week 4; 5 mg risperidone or 25 mg aripiprazole at week 6 and 6 mg risperidone or 30 mg aripiprazole at week 8. Study Psychiatrists will be able to increase faster if symptoms don't improve as well as decrease for side effects. These dose ranges conform with standard clinical practice and are within the FDA approved dosing ranges for schizophrenia, and schizoaffective disorder. Subjects advance in the risperidone titration schedule until they respond or develop dose-limiting side effects.
  Interventions: Drug: Risperidone or Aripiprazole (patients only)
- Healthy Volunteers: Healthy Volunteers will participate in MR imaging, Electroencephalogram , and cognitive testing.

INTERVENTIONS:
Drug: Risperidone or Aripiprazole (patients only) — Inpatients deemed eligible for the study, we be put on open-label risperidone
  Other Names: Risperidal; Aripiprazole
  Groups: Patients with Psychotic Disorders taking Risp. or Arip.

SUMMARY:
This is an observational neuroimaging treatment study. This study involves examining the neural circuitry of controlled treatment of patients presenting with a first-episode of psychosis with risperidone or aripiprazole. Patients who present for treatment of a first psychotic episode with a schizophrenia spectrum diagnosis and who are eligible to undergo treatment with either risperidone or aripiprazole will be offered participation in the study. Clinical ratings, neuropsychological testing, neuroimaging and EEG will be conducted at baseline. Additionally, subjects will undergo the same assessments at week 12 to determine treatment-related biomarkers. Clinical ratings, including neurocognitive testing, will be conducted by blinded raters at study visits during treatment. Healthy controls (N=50) will also be recruited and scanned twice (12-week interval) to control for effects of time and practice.

DETAILED DESCRIPTION:
In this proposed study, the study will examine treatment-related effects on functional brain circuitry in first episode schizophrenia. Converging lines of evidence suggest a key role for striatal disconnectivity in the pathophysiology of psychosis. The proposed study will utilize resting state functional magnetic resonance imaging (rs-fMRI), as well as fMRI tasks derived from the Research Domain Criteria (RDoC) framework, to: 1) develop and validate a prognostic biomarker to predict antipsychotic treatment response; and 2) to model the underlying neural circuitry changes associated with state changes in psychotic symptomatology. As a prognostic biomarker, a neuroimaging assay of striatal connectivity can potentially provide a clinically useful tool to advance the goal of precision medicine. As a longitudinal index of symptom change, our model can serve as an objective index against which to measure potential efficacy of newly developed antipsychotic treatments.

A large, well-characterized cohort of patients presenting with a first episode active psychosis (regardless of DSM diagnosis) will be recruited, along with matched controls. The study will utilize two well-validated fMRI tasks capturing two portions of the positive valence system: probabilistic category learning and reward responsiveness; these tasks are designed to interrogate dorsal and ventral corticostriatal circuits, respectively. The design will be longitudinal, with two scanning sessions performed for each patient: at baseline, and after 12 weeks of treatment. Treatment will be standardized across all patients to reduce potential confounds, and healthy controls will also be scanned at baseline and 12 weeks in order to control for effects of time and practice. Level of psychotic symptomatology (hallucinations, delusions, and thought disorder) will be measured at regular intervals using a comprehensive battery of rating scales. As secondary measures, electroencephalography (EEG) will be performed coinciding with neuroimaging on a subset of patients who provide consent. We will utilize Kaplan-Meier estimators and hierarchical linear modeling to examine the association of baseline striatal connectivity, and changes in connectivity over time, with clinical response of psychotic symptoms to antipsychotic treatment. Deliverables will include both baseline and longitudinal biomarkers that can subsequently be tested in broader, more heterogeneous populations of patients with psychosis.

ELIGIBILITY:
Patients

Inclusion Criteria:

1. current DSM-IV-defined diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, brief psychotic disorder, psychotic disorder NOS, bipolar I with psychotic features (acute manic or mixed episode), major depressive disorder with psychotic features as assessed using the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First et al, 1994);
2. does not meet DSM-IV criteria for a current substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, shared psychotic disorder, or a mood disorder without psychotic features;
3. current positive symptoms rated ≥4 (moderate) on one or more of these BPRS (Woerner et al., 1988) items: conceptual disorganization, grandiosity, hallucinatory behavior, unusual thought content;
4. is in a early phase of illness as defined by having taken antipsychotic medications for a cumulative lifetime period of 4 weeks or less,
5. age 15 to 40;
6. competent and willing to sign informed consent; and
7. for women, negative pregnancy test and agreement to use a medically accepted birth control method.

Exclusion Criteria:

1. serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain
2. any medical condition which requires treatment with a medication with psychotropic effects
3. significant risk of suicidal or homicidal behavior
4. cognitive or language limitations, or any other factor that would preclude subjects providing informed consent
5. medical contraindications to treatment with risperidone or aripiprazole monotherapy (e.g. neuroleptic malignant syndrome with prior risperidone exposure)
6. lack of response to a prior adequate trial of risperidone or aripiprazole

Healthy Volunteers

Inclusion

1. age 15 to 40
2. competent to sign informed consent

Exclusion

1. lifetime history of any mood disorder or any psychotic disorder as determined by clinical interview using the SCID-NP
2. MR imaging contraindications
3. neurologic conditions
4. any serious non-psychiatric disorder that could affect brain functioning
5. mental retardation

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Volunteers and Patients with Psychotic Disorders
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2016-07; Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
efficacy of risperidone or aripiprazole for psychotic symptoms | 12 weeks
  To examine the efficacious treatment of psychotic symptoms with either risperidone or aripiprazole measured by specific items on the Brief Psychiatric Rating Scale - conceptual disorganization, grandiosity, hallucinatory behavior, unusual thought content

SECONDARY OUTCOMES:
Relationship between efficacious treatment of psychotic symptoms and changes in functional connectivity of the striatum | 12 weeks
  To examine the relationship between efficacious treatment of psychotic symptoms (measured by the Brief Psychiatric Rating Scale) and changes in functional connectivity of the striatum, calculated from fMRI scans
Predicting treatment efficacy from baseline fMRI scans | 12 weeks
  To examine whether baseline fMRI scans can predict treatment efficacy which will be measured by the Brief Psychiatric Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Malhotra, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States